CLINICAL TRIAL: NCT05128604
Title: Introduction Of Endoscopic Ultrasound-Guided Gastroenterostomy Based On A Learning Protocol And Prospective Registry.
Brief Title: Endoscopic Ultrasound-Guided Gastroenterostomy Nationwide: Prospective Registry.
Acronym: GESICA
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Hospital Mutua de Terrassa (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital del Mar (Other); Germans Trias i Pujol Hospital (Other); Hospital Universitari de Girona Dr. Josep Trueta (Unknown); Hospital de Granollers (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario Virgen Macarena (Other); Hospital Universitario La Paz (Other); Hospital Universitario del Sureste (Other)
Responsible Party: Principal Investigator, Joan B Gornals, Principal Investigator, Director of Endoscopy Programme, Hospital Universitari de Bellvitge
Other Study IDs: GESICA
Record Dates: First submitted 2021-07-11; First posted 2021-11-22 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Endoscopic Surgical Procedure; Safety; Training
Keywords: endoscopic ultrasound; gastroenterostomy; lumen apposing stent
MeSH Terms: interventions — Gastroenterostomy; Endosonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Gastroenterostomy — Endoscopic ultrasound guided gastroenterostomy
  Other Names: Endoscopic ultrasound; Lumen apposing stent

SUMMARY:
This is project of help and support for the introduction of the GASTROENTEROANASTOMOSIS technique guided by ENDOSCOPIC -ULTRASOUND (EUS-GE) in centers in Catalonia, facilitating a teacher training.

The main objective is facilitate a safe introduction of the technique, limiting technical failures, and if necessary, support in rescue techniques.

The goal of this interventional study is to assess the impact of a teaching and on live-support model in the introduction of the gastroenteroanastomosis technique, evaluating its effects in safety and the learning curve.

regarding the results in safety and learning curve of for the introduction [type of study: observational study or clinical trial] is to [learn about, test, compare etc.] in [describe participant population/health conditions]. The main question[s] it aims to answer are:

* [question 1]
* [question 2] Participants will [describe the main tasks participants will be asked to do, treatments they'll be given and use bullets if it is more than 2 items]. If there is a comparison group: Researchers will compare [insert groups] to see if [insert effects].

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Gastric outlet obstruction (GOO) caused by passable /unpassable stenosis in the antrum-duodenal region, to malignant or non-malignant conditions
* Patient capable of understanding and signing informed consent form
* Patient understanding the type of study and complying with the follow-up of complementary tests during the study's duration

Exclusion Criteria:

* Massive ascites.
* Complete stenosis
* Failure to sign informed consent form
* Patients with intellectual handicap who are unable to understand the nature and possible consequences of the study, unless there is a competent legal representative
* Patients unable to adhere to subsequent follow-up requirements
* Severe coagulation disorder: INR > 1.5 not correctible with administration of plasma and/or platelets < 50,000/mm3

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with sympotmatic Gastric outlet obstruction (GOO) related to malignant or notn-malignant conditions.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2026-03-24 (Estimated); Study Completion 2026-09-24 (Estimated)

PRIMARY OUTCOMES:
Safety introduction of EUS-gastroenterostomy | 12 months
  To determine the safety of this interventional technique, measuring prospectively the adverse events and incidents after after a learning project for helping to introduce this technique.

SECONDARY OUTCOMES:
Learning curve | 12 months
  To assess the number of procedures related to a competence in the EUS-Gastroenterostomy

CONTACTS AND LOCATIONS:
Overall Officials: Joan B Gornals, MD, PhD, Principal Investigator — Hospital Universitari de Bellvitge - IDIBELL
Locations (6):
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol (Can Ruti), Badalona, Barcelona, Catalonia
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Catalonia
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Del Mar, Barcelona, Catalonia
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona, Catalonia

IPD SHARING:
Plan to Share IPD: Undecided